CLINICAL TRIAL: NCT02187978
Title: Comparison of Early Total Enteral Feeding (ETEF) Versus Conventional Enteral Feeding (CEF) in Stable Very Low Birth Weight (VLBW) Infants - A Randomized Controlled Trial
Brief Title: Early Total Enteral Feeding Versus Conventional Enteral Feeding in Stable Very Low Birth Weight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, Sushma Nangia, M.D., Dr Sushma Nangia, Professor of Pediatrics, Lady Hardinge Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LHMC/098/2012/ETEF
Record Dates: First submitted 2014-07-07; First posted 2014-07-11 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Nutrition of Preterm Infants
Keywords: Early total enteral feeding (ETEF); Conventional enteral feeding (CEF); VLBW infants; NEC; Preterm infants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early total enteral feeding (ETEF) (Experimental): Feeding will be initiated on D1 with 80ml/kg/day of expressed breast milk or LBW formula milk.
  No intravenous fluid will be provided. Feeds will be advanced till 150ml/kg/day is attained.
  Interventions: Other: Early total enteral feeding (ETEF)
- Conventional enteral feeding (CEF) (Active Comparator): Feeding will be initiated on D1of life with 20ml/kg of expressed breast milk or LBW formula milk.
  Remaining requirement as intravenous fluids. Feeds advanced by 20ml/kg/day for next 2 days and then 30ml/kg/day for the next three days until 150ml/kg/day is reached.
  Interventions: Other: Conventional enteral feeding (CEF)

INTERVENTIONS:
Other: Early total enteral feeding (ETEF) — In ETEF Group total required volume of fluid will be administered as oral feeds and no intravenous fluid will be given. Feeds will be started at 80 mL/kg and increased till 150ml/kg is attained.
  Arms: Early total enteral feeding (ETEF)
Other: Conventional enteral feeding (CEF) — CEF Group will receive some feed and some Intravenous fluids. Feeds will be slowly increased from 20 mL/kg on day 1 till full feeds 150ml/kg is attained on day 6 of life.
  Arms: Conventional enteral feeding (CEF)

SUMMARY:
The purpose of this study is to compare the effect of early total oral feeding versus conventional oral feeding in stable VLBW infants. In current clinical practice, the introduction of oral feeds for VLBW infants is often preceded by a period of fasting or minimal feeding because of fear of necrotizing enterocolitis (NEC). However, this may be associated with potential disadvantages and increased infectious and metabolic complications related to prolonged fasting and use of parenteral nutrition. The studies conducted till date have shown better outcomes and improved postnatal growth with early initiation and fast advancements of feeds. It is still unclear whether stable VLBW babies can tolerate total oral feeds on day 1 of life. No such study has been conducted on early total oral feeding but observational work in our unit has shown it to be safe without any increased incidence of feed intolerance or NEC. In view of the uncertainties regarding feeding protocols in VLBW infants all over the world, the investigators decided to assess the effect of early total enteral feeding in stable VLBW infants.

DETAILED DESCRIPTION:
Preterm VLBW infants often have negligible intrauterine reserves of nutrition along with a host of medical conditions postbirth including respiratory distress syndrome, hypoxia, hypotension, acidosis, infection and surgery. These conditions increase the metabolic energy requirements and nutrient needs of preterm babies. They require more specialised nutrition because of their faster growth rates; to correct the growth faltering post birth and to attain appropriate weight gain. Delayed postnatal growth due to inappropriate nutrition in early period leads to long term cognitive impairment and decreased school performance. Additional impediments to growth are high degree of biochemical and physiological immaturity of gastro intestinal tract with an immature immune system.

In current clinical practice, the introduction of progressive enteral feeds for preterm VLBW infants is often preceded by a period of enteral fasting or minimal enteral nutrition to decrease the incidence of NEC. However, there may also be potential disadvantages associated with delayed introduction of progressive enteral feeds. Gastrointestinal hormone secretion and motility is stimulated by enteral milk and hence delayed enteral feeding could diminish the functional adaptation of the gastrointestinal tract. In addition, 'starving' the gut may be harmful increasing susceptibility to infection due to impaired barrier function by intestinal epithelium. Parenteral nutrition (PN), though having an important role in early stabilization by allowing early calorie intake and preventing catabolism, is associated with significant risks of infectious and metabolic complications thereby increasing mortality and morbidity, prolonging hospital stay, and adversely affecting growth and development. As per recent literature reviews, enteral feeding has many advantages including appropriate intake of most nutrients. It also promotes growth and development of the gut and reduces the risk of infection. It is therefore important to establish enteral feeding as early as is safely possible. It has been argued that the risk of NEC should not be considered in isolation of these other potential clinical outcomes when determining feeding policies and practices for VLBW infants. A systematically conducted, randomized controlled trial is necessary to prove or refute the benefits of early total enteral feeding and nutrition. Hence the purpose of this prospective randomized controlled trial is to compare the benefits of early total enteral feeding over conventional enteral feeding in terms of attainment of full feeds, incidence of sepsis & NEC and duration of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Infants with gestational age between 28-34 weeks & hemodynamically stable preterm VLBW neonates (B Wt. 1000-1499g) defined as
* No asphyxia(not required resuscitation beyond initial steps)
* No significant respiratory distress at randomization (Not requiring respiratory support)
* No clinical evidence of shock at the time of randomization (not requiring vasopressor support)

Exclusion Criteria

* Major Congenital malformation
* Refusal of consent
* AREDF in utero

Ages: 30 Minutes to 120 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Day of attaining 150mL/Kg of enteral feeds | Till 45 days of age
  Full enteral feeds are defined as oral feeds at 150ml/Kg and sustaining it for 24 hrs

SECONDARY OUTCOMES:
Episodes of feed intolerance | Till 30 days of age or discharge whichever is earlier
  Feed intolerance defined as presence of 1 or more of the following
  * Vomiting >3 times during any 24 hr period
  * Any episode of bile/ blood stained vomiting
  * Abdominal girth (AG) increase > 2cm between feeds with pre feed gastric aspirate > 25% of pre feed volume (milk) or any amount hgic/bilious
  * Abdominal wall erythema
  * Gross blood in stools

OTHER OUTCOMES:
Incidence of Sepsis | Till 30 days of age or discharge whichever is earlier
  Incidence of suspect (Clinical setting with positive sepsis screen) and confirmed (Clinical setting with positive blood culture) sepsis in the two groups
Duration of Hospital Stay | Till 45 days of age
  The total duration of hospital stay till discharge alive from hospital will be calculated in completed number of days
Mean weight at one month of age | one month of age
  The difference in mean weight in grams at one month of age between the neonates of the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Sushma Nangia, MD,DM, Principal Investigator — Lady Hardinge Medical College & Kalawati Saran Children's Hospital
Locations (1):
- Lady Hardinge Medical College, New Delhi, National Capital Territory of Delhi, India